CLINICAL TRIAL: NCT04824690
Title: The Effect Of Immersive Virtual Reality Application On Anxiety, Pain And Family Satisfaction In The Perioperative Process Of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Aykut Turgut, Research Assistant, Abant Izzet Baysal University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2019_78
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Anxiety; Pain; Satisfaction
Keywords: Anxiety; Pain; Parental Satisfaction; Virtual Reality
MeSH Terms: conditions — Anxiety Disorders; Pain; Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): The virtual reality group watched a 1.5-minute VR video showing the operating theater and explaining the perioperative process. After the surgery, this group watched cartoons during the first standard nursing procedures after the effect of the anesthesia wore off.
  Interventions: Device: Virtual reality
- Control Group (No Intervention): The control group received conventional care and education regarding the perioperative process of surgery.

INTERVENTIONS:
Device: Virtual reality — Immersive virtual reality tour of the operating theatre before surgery and distraction methods both using VR headset
  Arms: Virtual Reality Group

SUMMARY:
An immersive virtual reality (VR) tour of the operating theater before surgery could reduce preoperative anxiety. The aims of this study were to analyze whether a preoperative virtual reality tour shows a reduction in anxiety in children and an increase in parental satisfaction.

DETAILED DESCRIPTION:
Children who will undergo surgery for the first time and their families were randomly allocated into the control or VR group. The control group received conventional education regarding the perioperative process of surgery. The VR group watched a 1.5-minute VR video showing the operating theater and explaining the perioperative process. The main finding was preoperative anxiety evaluated using the Children's State Anxiety (CSA) before surgery. Secondary findings included children's postoperative pain ratings using Wong-Baker Faces Pain Rating Scale and parental satisfaction scores using PedsQL Health Care Satisfaction Scale

ELIGIBILITY:
Inclusion Criteria:

* Children 4-10 years old
* ASA grade I or II
* General anesthesia
* Elective surgery

Exclusion Criteria:

* Children who have had previous surgery history
* Local anesthesia or emergency surgeries
* Premature or congenital disease history
* Having visual and hearing impairment
* Mental and developmental retardation
* Having a history of epilepsy and seizures
* Patients taking psychoactive drugs

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety assessed by the Children's State Anxiety (CAM-S) | This is measured right before the child goes into operating theatre / separating from his/her parents.
  The CAM-S scale is drawn to resemble a thermometer with a bulb at the bottom and horizontal lines at intervals going up to the top. Children are instructed to "Pretend that all of your worried or nervous feelings are in the bulb or bottom part of the thermometer. If you are a little bit worried or nervous, the feelings might come up in the thermometer just a little bit. If you are very, very worried or nervous, the feelings might go all the way to the top. Put a line on the thermometer showing how much worry or nervousness you feel. Min score : 0 & Max score : 10

SECONDARY OUTCOMES:
Postoperative Pain assessed by the Wong-Baker Faces Pain Rating Scale | This is measured immediately after the surgery.
  The scale is used around the world with people ages 3 and older. Min score : 0 & Max score : 5
Parental Satisfaction assessed by PedsQL Health Care Satisfaction Scale | This is measured immediately after the intervention.
  Parents answered the following scale questions by indicating how satisfied they are with the services provided to them and their children. Min score : 0 & Max score : 100
Postoperative anxiety assessed by the Children's State Anxiety (CAM-S) | This is measured immediately after the surgery.
  The CAM-S scale is drawn to resemble a thermometer with a bulb at the bottom and horizontal lines at intervals going up to the top. Children are instructed to "Pretend that all of your worried or nervous feelings are in the bulb or bottom part of the thermometer. If you are a little bit worried or nervous, the feelings might come up in the thermometer just a little bit. If you are very, very worried or nervous, the feelings might go all the way to the top. Put a line on the thermometer showing how much worry or nervousness you feel. Min score : 0 & Max score : 10

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No